CLINICAL TRIAL: NCT00434603
Title: Expressive Arts as a Social and Community Integration Tool for Adolescents With Acquired Brain Injury: "I Want to Thrive, Not Just Survive!"
Brief Title: Expressive Arts as a Social and Community Integration Tool for Youth Recovering From Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Michelle Keightley, Assistant Professor, University of Toronto
Other Study IDs: 001
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Expressive Arts--Theatre Skills Training Program — The experimental intervention was an intensive theatre skills training program. The group of adolescent participants recovering from ABI met daily for four hours over a period of 4 weeks. During this 4 hour period, regular breaks were scheduled to provide the participants with a mental and physical break from therapy. Theatre training included voice work, breathing, movement, physical warm-up, character development, script analysis, writing skills, three-dimensional awareness, group dynamics, story development, mask work and clowning among others.

SUMMARY:
This study utilizes a novel technique-expressive arts therapy-to facilitate social integration for youth recovering from acquired brain injury (ABI). Expressive arts therapy is defined as the use of the arts and artistic media to explore psychological aspects of life. An expressive art (also referred to as 'creative arts' or even just 'arts') encompasses drama, music, art (visual arts such as painting, sculpture etc) and dance/movement. It has great potential to improve community integration for youth recovering from ABI, through facilitating skills required for successful social communication and social cognition. It is hypothesized to improve social and emotional functioning compared to a less structured creative arts program. It is expected that a combination of directed group activities and self-reflection within a creative learning context will improve emotional awareness and social and community integration to a greater degree than a non-expressive creative arts therapy group, in youth who have suffered an ABIAs community integration enables meaningful and productive occupational engagement, enabling opportunities for occupational engagement through increased community integration would greatly enhance the quality of life of adolescents with ABI.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months post injury
* Difficulties in social and emotional functioning
* Entering Grades 10 and 11 in 2007
* English fluency

Exclusion Criteria:

* Extreme behaviour, mood and cognitive disturbance

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Youth recovering from acquired brain injury
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Keightley, Principal Investigator — University of Toronto